CLINICAL TRIAL: NCT02076126
Title: Spectroscopic-chemometric Determination of Lecithin-sphingomyelin Ratio in Gastric Aspirates and Secretion From Hypopharynx at Birth, in Relation to Development of RDS
Brief Title: Determination of Lung Maturity and Prediction of RDS at Birth
Status: Completed | Type: Observational
Sponsor: Henrik Axel Verder (Other)
Collaborators: Holbaek Sygehus (Other); Aalborg University Hospital (Other); Odense University Hospital (Other); Aarhus University Hospital Skejby (Other); Kolding Sygehus (Other); Copenhagen University Hospital at Herlev (Other); Rigshospitalet, Denmark (Other); Hvidovre University Hospital (Other); Naestved Hospital (Other); University Hospital, Linkoeping (Other); Skane University Hospital (Other)
Responsible Party: Sponsor-Investigator, Henrik Axel Verder, Professor DMSc, Holbaek Sygehus
Organization: Holbaek Sygehus (Other)
Other Study IDs: Holb.SJ-384
Record Dates: First submitted 2014-02-28; First posted 2014-03-03 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: RDS; Premature Birth
Keywords: Lung maturity; RDS; Prematurity; Lecithin-sphingomyelin ratio; Spectroscopy; Chemometrics
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Gastric- and hypopharyngeal secretions
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Gastric aspirate: L/S ratio on the gastric aspirates are retrospectively compared with the possible development of RDS
- Hypopharyngeal secretion: L/S ratio on the hypopharyngeal secretions are retrospectively compared with the possible development of RDS

SUMMARY:
The overall objective is to identify quickly after birth the preterm infants who will develop respiratory distress syndrome (RDS) for the purpose of treating them as early as possible with surfactant, to reduce, and if possible, to avoid sequelae, including long-term oxygen treatment.

We have therefore developed a quick test, which we believe will be ideal for this type of diagnostics, and will now test the method in a preclinical trial.

DETAILED DESCRIPTION:
In at least 135 preterm infants with gestational age 24-32 weeks we will collect gastric aspirate and hypopharyngeal secretion. The infants are stratified into three groups: gestational age 24-25 weeks, 26-29 weeks and 30-31 weeks.

The aspirates will be frozen at -20 centigrade and lecithin-sphingomyelin ratio (L/S) will be analysed retrospectively using Fourier Transform Infrared Spectroscopy.

The infants will be monitored for the first five days with regard to possible development of RDS.

Clinical and biochemical data will be compared retrospectively.

There a no intervention procedures.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with gestational ages of 24 (24+0) to 32 (31+6) weeks.
* Age < ½ hour

Exclusion Criteria:

* Lack of informed consent
* lack of aspirate

Ages: 1 Minute to 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 135 preterm infants with gestational age 24-32 weeks (24+0 to 31+6)
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
RDS | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Verder, Professor MD, Principal Investigator — Holbaek Hospital
Locations (1):
- Holbaek Sygehus, Holbæk, Denmark